CLINICAL TRIAL: NCT07205913
Title: Gut Microbiota, Diet-INDuced Obesity and Type 2 Diabetes in New Caledonia - MIND
Acronym: MIND
Status: Not yet recruiting | Type: Observational
Sponsor: Institut Pasteur (Industry)
Collaborators: RIKEN Center for Integrative Medical Sciences (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2025-020; 2025-A01257-42 (Other: ID-RCB)
Record Dates: First submitted 2025-09-25; First posted 2025-10-03 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Diabetes Mellitus, Type 2; Obesity
Keywords: microbiota; New Caledonia; metabolic diseases
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity; Metabolic Diseases | interventions — Blood Specimen Collection; Defecation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood sample Urine stools
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Obese group with a BMI ≥30 with type 2 diabetes
  Interventions: Other: 25 ml blood sample; Other: Urine sample; Other: Stools
- Obese group with a BMI ≥30 without any type of diabetes
  Interventions: Other: 25 ml blood sample; Other: Urine sample; Other: Stools
- Control group of participants considered as "metabolically healthy"
  Interventions: Other: Urine sample; Other: Stools; Other: 40 ml blood sample

INTERVENTIONS:
Other: 25 ml blood sample — A 25-ml blood sample
  Groups: Obese group with a BMI ≥30 with type 2 diabetes; Obese group with a BMI ≥30 without any type of diabetes
Other: Urine sample — A 10-ml urine sample
Other: Stools — 10-g stools
Other: 40 ml blood sample — A 40-ml blood sample
  Groups: Control group of participants considered as "metabolically healthy"

SUMMARY:
In recent years, the global rise in obesity and type 2 diabetes has become a major public health issue. In New Caledonia, 38% of the adult population has a body mass index ≥30. At the same time, the prevalence of type 2 diabetes continues to rise steadily. The burden of these diseases does not affect communities uniformly. While known factors such as diet, physical activity, and socioeconomic conditions play a role, studies have demonstrated the involvement of the gut microbiota in the development of metabolic disorders, particularly obesity and insulin resistance. However, this area remains largely unexplored in New Caledonia and the Pacific.

DETAILED DESCRIPTION:
The goal of the study is to describe and characterize the gut microbiota and fecal metabolome of participants and study the relationships between microbiota composition and bioclinical parameters in participants with different metabolic states, ranging from "metabolically healthy" to severe obesity with and without type 2 diabetes.

To achieve this goal, adults in New Caledonia divided in 3 groups

1. Obese group with a BMI ≥ 30 with type 2 diabetes,
2. Obese group with a BMI ≥ 30 without any type of diabetes,
3. Control group of participants with a BMI between 18.5 and 24.9 kg/m2 and without any type of diabetes.

will be recruited. Blood, urine, and stool samples will be collected from participants. A questionnaire to collect sociodemographic characteristics as well as behaviors and lifestyle habits related to diet, physical activity, and psychological health.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 60 years.
* Ability to understand and provide informed consent.
* Ability and willingness to meet the required schedule and study interventions.
* Willingness to share their community belonging
* Benefit from a social security system.

For obese and diabetic patients :

* IMC ≥ 30 kg/m² with type 2 diabetes
* Fasting plasma glucose (FPG) ≥7 mM (=1.26g/l) or
* Patients with HbA1c ≥ 6.5% (48 mmol/mol)
* All stages of albuminuria For obese patients without type 2 diabetes
* IMC ≥ 30 kg/m²
* Weight stable for at least 2 months
* Patients with normal glucose tolerance (NGT), impaired glucose tolerance (IGT) and/or impaired fasting glucose (IFG) and an HbA1c < 6.5 %
* No treatment (diabetic or weight loss)
* Match age (±5years), sex and self-reported community to the patients from the1 group.

For control group :

* BMI between 18.5-24.9 kg/m²
* Match age (±5years), sex and self-reported community to the patients from the 1 and 2 groups.
* Participants with normal glucose tolerance (NGT), impaired glucose tolerance (IGT) and/or impaired fasting glucose (IFG) and an HbA1c < 6.5 %

Exclusion Criteria:

All participants :

* Treatment that may alter gastrointestinal motor function, acidity, microbial population, or immunosuppressants
* Altered anatomy of the esophagus, stomach, small intestine, or large intestine due to gastrointestinal surgery (except appendectomy or cholecystectomy)
* Chronic or acute inflammatory bowel disease or infections
* Abdominal or pelvic radiation therapy or abdominal cancer, colorectal cancer
* Dysphagia, eosinophilic esophagitis, esophageal stricture, or other swallowing disorders
* Organ transplantation and patients receiving immunosuppressive therapy
* Severe renal failure and/or patients undergoing dialysis
* Cardiovascular, endocrine, renal, or other chronic disease that may affect motility.
* Preparation for colon cleansing within the last month
* < 3 bowel movements per week
* Women who are pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults living in New Caledonia who are obese with or without type 2 diabetes or healthy
Sampling Method: Probability Sample
Enrollment: 270 (Estimated)
Dates: Start 2025-11-15 (Estimated); Primary Completion 2026-11-15 (Estimated); Study Completion 2026-11-15 (Estimated)

PRIMARY OUTCOMES:
Describe and characterise the faecal microbiota of patients to investigate the relationships between microbiota composition with bioclinical parameters | 6 years
  Microbiota will be analysed through 16S rRNA gene sequencing as well as shotgun metagenomic sequencing of the different samples obtained from the faecal sample
Describe and characterise the faecal microbiota and metabolome of patients to investigate the relationships between microbiota composition with bioclinical parameters | 6 years
  microbiome and metabolites from collected human fecal samples will be analyzed using a standardized extraction protocol designed for Liquid chromatography-mass spectrometry (LC/MS)-based metabolomics to detect short-chain fatty acids and bile acids,…. which are mainly produced by bacteriasequencing of the different samples obtained from the faecal sample.